CLINICAL TRIAL: NCT03887884
Title: Randomized, Multi-center, Open-label, Crossover Pharmacokinetic Study of CVT-301 (Levodopa Inhalation Powder) and an Oral Dose of Carbidopa/Levodopa CD/LD Under Fed Conditions in Patients With Parkinson's Disease
Brief Title: Pharmacokinetic Study of CVT-301 (Levodopa Inhalation Powder)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acorda Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CVT-301-012
Record Dates: First submitted 2019-03-01; First posted 2019-03-25 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-08

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — carbidopa, levodopa drug combination

STUDY DESIGN:
Intervention Model Description: It is a 2-way crossover Pharmacokinetic (PK) evaluation of a single inhaled dose of CVT-301 84 mg and a single oral dose of Carbidopa/levodopa (CD/LD) 25 mg/100 mg (Sinemet®) under fed conditions in Parkinson's Disease patients who regularly take CD/LD.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CVT-301 (Experimental): Single inhaled dose of CVT-301 84 mg
  Interventions: Drug: CVT-301
- Sinemet (Active Comparator): Single oral dose of Carbidopa/Levodopa 25 mg/100 mg
  Interventions: Drug: Sinemet

INTERVENTIONS:
Drug: CVT-301 — Levodopa Inhalation Powder
  Arms: CVT-301
Drug: Sinemet — Single oral dose of Carbidopa/Levodopa 25 mg/100 mg
  Arms: Sinemet

SUMMARY:
This study will be an open-label, randomized, multi-center, 2-way crossover Pharmacokinetic PK evaluation of a single inhaled dose of CVT-301 84 mg and a single oral dose of carbidopa/levodopa CD/LD 25 mg/100 mg (Sinemet®) under fed conditions in Parkinson's Disease (PD) patients who regularly take CD/LD.

DETAILED DESCRIPTION:
The study duration includes a screening period followed by an overnight stay in the center (4 days, 3 nights) to complete 2 treatments, including a 48-hour interval between the treatments, and a follow-up phone call 1-2 days after discharge from the center.

On each of two treatment days, subjects will consume a standard high fat meal and then receive either (A) a single inhaled dose of CVT-301 or (B) a single dose of oral CD/LD followed by Pharmacokinetic (PK) sampling for 4 hours. A crossover design will be used such that each subject receives both Treatment A and Treatment B over the 2 treatment days, randomized 1:1 to the treatment sequence AB or BA.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 30 and 85 years, inclusive.
* Have idiopathic PD (i.e., not induced by drugs or other diseases) as defined by fulfilling Steps 1 and 2 of the United Kingdom (UK) Brain Bank criteria, diagnosed after the age of 30 years.
* Classified as Stage 1 to 3 (in the ON state) on the modified Hoehn and Yahr scale for staging of PD severity.
* Stable on other non levodopa PD medications for at least 4 weeks prior to the Screening Visit.
* Subjects must have normal cognition as confirmed by a score of ≥ 25 on the Mini Mental State Examination (MMSE), performed in the ON state.
* Forced expiratory volume in one second (FEV1) ≥60% of predicted for race, age, sex, and height and FEV1/FVC (forced vital capacity) ratio ≥70%.
* Body Mass Index (BMI) between 18 - 32 kg/m2, inclusive.

Exclusion Criteria:

* Any flu-like syndrome or other respiratory infections within 2 weeks prior to the Screening Visit.
* Chronic obstructive pulmonary disease (COPD), asthma, or other chronic respiratory disease within the last 5 years.
* History of any cancer in the past 5 years with the exception of successfully treated basal cell carcinoma.
* Narrow angle glaucoma or a history of peptic ulcer disease less than 1 year prior to screening.
* Previous surgery for PD (including but not limited to deep brain stimulation or cell transplantation).
* Current use of nicotine patch or tobacco-containing products including cigarettes, electronic cigarettes, cigars, chewing tobacco, pipe tobacco or snuff or use within 4 weeks prior to the Screening Visit, or expected use during the study.
* Marijuana smoking within 4 weeks prior to the Screening Visit, or expected smoking/inhalation during the study.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration of a single inhaled dose of CVT-301 84 mg and an oral dose of CD/LD 25 mg/100 mg (carbidopa/levodopa) in patients with Parkinson's disease. | 4 days, 3 nights
  Maximum observed plasma drug concentration (Cmax) of a single inhaled dose of CVT-301 84 mg and an oral dose of CD/LD 25 mg/100 mg in patients with Parkinson's disease (PD) in a fed state.
Total plasma concentration of a single inhaled dose of CVT-301 84 mg and an oral dose of CD/LD 25 mg/100 mg (carbidopa/levodopa) in patients with Parkinson's disease. | 4 days, 3 nights
  Area under the plasma concentration curve from time 0 to the concentration at 4 hours (AUCo-4h) of a single inhaled dose of CVT-301 84 mg and an oral dose of CD/LD 25 mg/100 mg in patients with Parkinson's disease (PD) in a fed state.
Terminal half-life of a single inhaled dose of CVT-30184 mg and an oral dose of CD/LD 25 mg/100 mg (carbidopa/levodopa) in patients with Parkinson's disease. | 4 days, 3 nights
  Terminal half-life (t1/2)of a single inhaled dose of CVT-30184 and an oral dose of CD/LD 25 mg/100 mg in patients with Parkinson's disease (PD) in a fed state.
Time to maximum observed plasma drug concentration of a single inhaled dose of CVT-301 84 mg and an oral dose of CD/LD 25 mg/100 mg (carbidopa/levodopa) in patients with Parkinson's disease. | 4 days, 3 nights
  Time to maximum observed plasma drug concentration (Tmax) of a single inhaled dose of CVT-301 84 mg and an oral dose of CD/LD 25 mg/100 mg in patients with Parkinson's disease (PD) in a fed state.

SECONDARY OUTCOMES:
Columbia-Suicide Severity Rating Scale (C-SSRS). | 4 days, 3 nights
  To evaluate the safety and tolerability of a single inhaled dose of CVT-301 84 mg and an oral dose of CD/LD 25/100 mg) under fed conditions in PD patients using the Columbia-Suicide Severity Rating Scale (C-SSRS). The (C-SSRS) is an assessment tool that evaluates suicidal ideation and behavior. Scale range: Yes or No response to 10 questions, with minimum to maximum range of 0 to 10. Lower score represents better outcomes. Subscales not applicable.
Incidence of adverse events. | 4 days, 3 nights
  To evaluate the safety and tolerability of a single inhaled dose of CVT-301 84 mg and an oral dose of CD/LD 25/100 mg) under fed conditions in PD patients by accessing adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Oh, MD, Study Director — Acorda Therapeutics
Locations (5):
- United States (5):
  - Acorda Site #1003, Long Beach, California
  - Acorda Site #1005, Hallandale, Florida
  - Acorda Site #1002, Orlando, Florida
  - Acorda Site #1004, Atlanta, Georgia
  - Acorda Site #1001, Farmington Hills, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Safirstein BE, Ellenbogen A, Zhao P, Henney HR 3rd, Kegler-Ebo DM, Oh C. Pharmacokinetics of Inhaled Levodopa Administered With Oral Carbidopa in the Fed State in Patients With Parkinson's Disease. Clin Ther. 2020 Jun;42(6):1034-1046. doi: 10.1016/j.clinthera.2020.04.004. Epub 2020 May 29. PMID 32482490